CLINICAL TRIAL: NCT00375518
Title: Double-Blind Study of Atorvastatin Versus Placebo to Reduce Cardiopulmonary Complications After Thoracic Surgery
Brief Title: Study of Atorvastatin Versus Placebo to Reduce Cardiopulmonary Complications After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 06-079
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Thoracic Surgery
Keywords: Thoracic Surgery; Cardiopulmonary complications; Atorvastatin
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40 mg once a day beginning 7 days before the operation. Surgical procedures will be as planned and unaffected by this study. Starting from the day after surgery, patients will be given their study drug for an additional 7 days.
  Arms: 1
Drug: Placebo — Placebo given beginning 7 days before the operation. Starting from the day after surgery, patients will be given their study drug for an additional 7 days.
  Arms: 2

SUMMARY:
This study will compare atorvastatin (Lipitor) with a placebo (inactive pill) to see if this drug reduces heart rhythm abnormalities (arrhythmias) or lung inflammation after thoracic surgery. Preliminary results suggest that cholesterol lowering drugs (statins) may reduce problems after surgery such as arrhythmias or lung inflammation which may be serious. This study will be randomized and double blind, meaning that patients are placed in groups purely by chance, like flipping a coin. Neither the patient or doctor will know which group the patient is in.

DETAILED DESCRIPTION:
Hypothesis: Statins attenuate perioperative inflammatory and oxidative mechanisms that contribute to the initiation and severity of cardiopulmonary complications after thoracic surgery.

Aim 1. To determine whether prophylactic administration of atorvastatin attenuates the inflammatory and oxidative response to surgery and significantly reduces the composite risk of cardiovascular morbidity (atrial fibrillation (AF), acute coronary syndrome, myocardial infarction (MI), cerebrovascular accident (CVA), pulmonary embolism) and mortality within 30 days after thoracic surgery.

Aim 2. To explore whether prophylactic administration of atorvastatin attenuates the inflammatory and oxidative (CRP, IL-6, TNF, and MPO) response to surgery and significantly reduces the overall risk of pulmonary complications (atelectasis, pneumonia, pneumonitis, acute respiratory failure) after thoracic surgery.

Aim 3. To explore the association of single nucleotide polymorphism (SNP) changes in genes linked to atrial fibrillation and inflammatory markers and development of pulmonary morbidity after thoracic surgery.

Aim 4. To explore whether an imbalance between metalloproteinase (MMP)-1 and its inhibitor (TIMP) is associated with postoperative atrial fibrillation risk and/or development of pulmonary morbidity after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 yr. scheduled for anatomic lung resection (segmentectomy, lingulectomy, possible or definite lobectomy, bilobectomy, pneumonectomy or extrapleural pneumonectomy) with or without chest wall resection or limited resection
* Patients with regular cardiac rhythm
* Patients able to take oral capsules
* Patients capable of providing written, informed consent
* Patients without known hepatic or kidney disease

Exclusion Criteria:

* Patients already taking any statin, gemfibrozil (Lopid), or ezetimibe (Zetia)
* Hypersensitivity to atorvastatin
* Chronic atrial fibrillation
* Patients already taking class Ic or III antiarrhythmic drugs
* Known pregnancy a urine pregnancy test will be given to women of childbearing age
* Known history of active hepatic disease or known hepatic insufficiency
* Known history of active kidney disease or insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Amar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- [Derived] Amar D, Park B, Zhang H, Shi W, Fleisher M, Thaler HT, Rusch VW. Beneficial effects of perioperative statins for major pulmonary resection. J Thorac Cardiovasc Surg. 2015 Jun;149(6):1532-8. doi: 10.1016/j.jtcvs.2014.12.016. Epub 2014 Dec 18. PMID 25623903
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 80 | 82
Completed | 72 | 65
Not Completed | 8 | 17
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Patient Not Treated | 6 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 46 | 83
  >=65 years | 43 | 36 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Determine the Postoperative Complications Found in Each Group
Description: To determine whether one week of preventive therapy with atorvastatin prior to surgery and one week after surgery reduced the composite rate of cardiovascular morbidity when compared to placebo.
Time Frame: one week (minimum of 5 days) before surgery and continued for one week (minimum of 5 days) after surgery
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 72 | 65
participants
  With Post Operative Complications | 16 | 8
  Without Post Operative Complications | 56 | 57

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/82
Other Adverse Events (participants affected / at risk) | 31/80 | 33/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=80) | Placebo (N=82)
Adult Respiratory Distress Synd (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=80) | Placebo (N=82)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 15 (15) | 17 (17)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 12 (12) | 20 (20)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes